CLINICAL TRIAL: NCT06562595
Title: What is the Optimal Training Model for Cervical Awareness?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Celal Akdemir, Department of Gynecologic Oncology, Principal Investigator, Izmir City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ISH
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: HPV Infection; Cervical Cancer; Cervical Dysplasia
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: The training methods employed comprise four arms:
  1. Video-based training,
  2. Classical lecturing,
  3. Brochure,
  4. Voice recording (Radio broadcast).
Who Masked: Participant
Masking Description: The participant will be randomly assigned to one of the four experimental groups by a computerised randomisation software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Video Assisted (Experimental): Those participants who are automatically assigned to the video training arm will be required to complete a 25-point initial assessment, after which they will be presented with a video. Subsequently, the same test will be administered once more, and the initial and subsequent scores of the participant will be recorded in the case report form.
  Interventions: Behavioral: Education Intervention
- Classical Lectures (Experimental): The initial assessment, comprising 25 items, will be administered to participants who have been randomly assigned to the control group. This group will be invited to attend a seminar at our clinic, during which a PowerPoint presentation will be delivered. Following the conclusion of the presentation, the same assessment will be repeated, and the participant's initial and second scores will be recorded in the case report form.
  Interventions: Behavioral: Education Intervention
- Brochure (Experimental): Those participants who are automatically assigned to the brochure arm will be required to complete a 25-point initial test. Participants assigned to this arm will receive a web-based brochure on HPV and smear information (via free messaging services). At the conclusion of the brochure review, the same test will be administered again, and the participant's initial and second scores will be recorded in the case report form.
  Interventions: Behavioral: Education Intervention
- Sound Recording (Radio Broadcast) (Experimental): Participants who have been automatically assigned to the Sound Recording (Radio Broadcast) arm will be required to complete a 25-point initial assessment. This assessment will be administered via a web-based platform, accessible through free messaging services. Following the completion of the Sound Recording (Radio Broadcast), the same assessment will be repeated. The initial and second scores will then be recorded in the case report form.
  Interventions: Behavioral: Education Intervention

INTERVENTIONS:
Behavioral: Education Intervention — Training will be provided to the participants, with the objective of determining the most accurate training method on HPV and cervical awareness.

SUMMARY:
Cervical cancer represents the fourth most prevalent malignant disease and the fourth leading cause of mortality among women on a global scale. Despite screening and preventive vaccination efforts, cervical cancer remains a significant cause of morbidity and mortality in low- and middle-income countries.

DETAILED DESCRIPTION:
A number of studies have been conducted with the aim of raising awareness about HPV and cervical cancer. However, there is currently no evidence-based consensus on the most effective method of education. The objective of this study is to identify the optimal training method by conducting a randomised controlled trial among healthcare professionals. The training methods under consideration are as follows: 1) Video-based training, 2) Classical lecture training, 3) Brochure, 4) Audio recording (Radio broadcast).

Prior to the commencement of the designated training methods, participants will be required to complete a web-based pre-test. Subsequent to this, the system will automatically assign each participant to a training intervention. Upon completion of the training programme, participants will be required to undertake a second test, the results of which will inform the selection of the most effective training method.

This study will be conducted separately in several distinct healthcare professional groups. Each randomized controlled trial will include 400 participants.

Planned groups include:

Public health nurses

Medical doctors

Medical interns

Midwives

The objective is to identify the most effective educational intervention for improving awareness of HPV and cervical cancer prevention within each group.

ELIGIBILITY:
Inclusion Criteria:

Being over 18 and under 40

* Female doctors, female nurses and female health technicians
* Working in our hospital
* Having sufficient mental capacity
* Not having a visual or auditory disability
* Volunteering to participate in the study

Exclusion Criteria:

* Under 18 and over 40
* Not being a healthcare worker
* Not having enough mental capacity
* Having a visual or auditory disability
* Patients who did not volunteer to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Test Score, Pre-Training | After completion of the 25-item assessment tests (first and second test) and training, an average of 1 month.
  Participants will first take a test where they will receive a maximum of 25 points and a minimum of 0 points. Then the participants will be automatically assigned to one of the 4 training models, then the trainings will be given and the same test will be applied to the participants again.
  By looking at the second test and first test scores, it will be determined which training model increases the participant's score more. Thus, we will be able to understand which form of education increases HPV and cervical awareness in our society.
Test Score, Post-Training | After completion of the 25-item assessment tests (first and second test) and training, an average of 1 month.
  Participants will first take a test where they will receive a maximum of 25 points and a minimum of 0 points. Then the participants will be automatically assigned to one of the 4 training models, then the trainings will be given and the same test will be applied to the participants again.
  By looking at the second test and first test scores, it will be determined which training model increases the participant's score more. Thus, we will be able to understand which form of education increases HPV and cervical awareness in our society.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir City Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
What is the most efficacious method of disseminating information about the human papilloma virus (HPV) and cervical cancer awareness?
Supporting Information: Study Protocol